CLINICAL TRIAL: NCT00734994
Title: Pilot Study of External Hyperthermia and Intravesical Mitomycin-C To Treat Recurrent Bladder Cancer After Resection and Standard Adjuvant Therapy
Brief Title: Mitomycin C With Hyperthermia and Intravesical Mitomycin C to Treat Recurrent Bladder Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mark Dewhirst (Other)
Responsible Party: Sponsor-Investigator, Mark Dewhirst, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003239
Record Dates: First submitted 2008-05-04; First posted 2008-08-14 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Transitional Cell Carcinoma of Bladder; Superficial Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperthermia system, Mitomycin C (Experimental): Pilot study single arm study to test the safety, tolerability and clinical benefit of regional hyperthermia and mitomycin-C intravesical chemotherapy to treat non-invasive Transitional Cell carcinoma (TCC) of the bladder that has recurred after standard resection and adjuvant therapy.
  Interventions: Device: Hyperthermia System; Drug: Mitomycin C

INTERVENTIONS:
Device: Hyperthermia System — Hyperthermia applied to heat the bladder to a temperature of 42 degrees Celsius for 40-60 minutes concurrent with mitomycin Treatment Schedule: 6 Weekly Sessions (Induction) followed by 4 Monthly Sessions (Maintenance) until documented second recurrence
  Other Names: BSD 2000 Hyperthermia system
Drug: Mitomycin C — 40 mg in 40 ml sterile water instilled into bladder
  Other Names: Mutamycin

SUMMARY:
Hypothesis: In selected patients external hyperthermia will be used in combination with intravesical Mitomycin-C (MMC) to treat recurrent transitional cell carcinoma (TCC) of the bladder after local resection and standard adjuvant therapy and thus prevent or delay recurrence and the need for radical cystectomy.

DETAILED DESCRIPTION:
It is well established that tumor cells are sensitive to heat and when combined with a chemotherapeutic agent, drug uptake and intracellular distribution of drug within malignant cells is improved due to increased cellular permeability. Further, hyperthermia inhibits deoxyribonucleic acid (DNA) repair as a result of increased reaction between DNA and chemotherapy. By heating bladder tissue and accelerating the necessary series of reactions to link agents such as mitomycin C to cell DNA, this effect may be optimized. Depending on the extent of resection (and location, size, and depth of invasion of remaining tumor) after transurethral resection of the bladder tumor(TURBT), recommended adjuvant therapy consists of intravesical chemotherapy. MMC has been studied at doses as high as 80 mg without producing significant or irreversible side effects. The most commonly used dose of mitomycin is 40 mg.2

This pilot study proposes to use Mitomycin C at a dose of 40 mg in conjunction with deep hyperthermia to enhance the effect intravesical chemotherapy as second-line treatment of recurrent TCC (Stage Ta, T1, or Tis) of the bladder after surgical resection and standard adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-muscle invasive transitional cell carcinoma (TCC) of the bladder (Ta, T1, Tis) recurrent after initial surgery and at least one round of adjuvant treatment (i.e. 6 weeks of intravesical biological therapy with Bacillus Calmette Guerin (BCG) solution); or
* An inability to tolerate BCG
* Age > 18
* Eastern Cooperative Oncology Group(ECOG) Performance Status 0-2
* Laboratory tests performed within 14 days of study enrollment:

  * Leukocytes ≥ 3,200, Absolute Neutrophil count ≥ 1,500, Platelets ≥ 100,000
  * Hemoglobin ≥ 9.0 gm/dL, Total bilirubin ≤ institution upper limit of normal *(ULN), Asparate Aminotransferase(AST) and Alanine Aminotransferase(ALT) ≤ 2.5 times ULN, Alkaline phosphatase ≤ 2.5 times ULN
  * Creatinine ≤ 1.5 times ULN
* Women of child bearing potential must have a negative pregnancy test
* If post-menopausal - Amenorrhea for ≥ 12 months

Exclusion Criteria:

* Pregnancy or breastfeeding
* Muscle invasive disease (T2-T4)
* Prior radiation to the pelvis
* Peripheral neuropathy (any grade)
* Thrombocytopenia, coagulation disorder or an increase in bleeding tendency due to other causes
* Known bladder fistula
* Hypersensitive or idiosyncratic reaction to mitomycin-C or its components in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zelko Vujaskovic, MD, Principal Investigator — Duke University; Brant A Inman, MD, MS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Juang T, Stauffer PR, Craciunescu OA, Maccarini PF, Yuan Y, Das SK, Dewhirst MW, Inman BA, Vujaskovic Z. Thermal dosimetry characteristics of deep regional heating of non-muscle invasive bladder cancer. Int J Hyperthermia. 2014 May;30(3):176-83. doi: 10.3109/02656736.2014.898338. Epub 2014 Mar 26. PMID 24669804
- [Background] Yuan Y, Cheng KS, Craciunescu OI, Stauffer PR, Maccarini PF, Arunachalam K, Vujaskovic Z, Dewhirst MW, Das SK. Utility of treatment planning for thermochemotherapy treatment of nonmuscle invasive bladder carcinoma. Med Phys. 2012 Mar;39(3):1170-81. doi: 10.1118/1.3679839. PMID 22380348
- [Result] Inman BA, Stauffer PR, Craciunescu OA, Maccarini PF, Dewhirst MW, Vujaskovic Z. A pilot clinical trial of intravesical mitomycin-C and external deep pelvic hyperthermia for non-muscle-invasive bladder cancer. Int J Hyperthermia. 2014 May;30(3):171-5. doi: 10.3109/02656736.2014.882021. Epub 2014 Feb 3. PMID 24490762

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 09/2008-09/2010 Location: Urology and Radiation Oncology Clinics
Groups:
- Mitomycin C With Hyperthermia and Recurrent Bladder Cancer: Mitomycin C with Hyperthermia to Treat Recurrent Bladder Cancer
Period: Overall Study
Arm/Group | Mitomycin C With Hyperthermia and Recurrent Bladder Cancer
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Mitomycin C With Hyperthermia: Mitomycin C and Hyperthermia
Arm/Group | Mitomycin C With Hyperthermia
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Secondary Outcome: Median Recurrence Free-survival
Description: Time to first recurrence of cancer in the bladder.
Time Frame: Median follow-up 3.18 years
Population: Entire cohort
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Hyperthermia System, Mitomycin C
Number analyzed (Participants) | 15
Months | 15.4 [12.2 to NA] — Confidence interval not calculable due to insufficient number of participants.

2. Primary Outcome: Safety and Tolerability
Description: Number of patient treatments stopped due to safety concerns or treatment intolerability. All events below are grade 1/2 toxicity. No grade 3-5 toxicity was observed.
Time Frame: During Treatment Phase average 6 weeks
Measure: Number; unit: Grade 1/2 event count (no grade 3+)
Units Other Than Participants: Hyperthermia Treatments
Arm/Group | Mitomycin C With Hyperthermia
Number analyzed (Participants) | 15
Number analyzed (Hyperthermia Treatments) | 132
Grade 1/2 event count (no grade 3+)
  Abdominal pain | 5
  Fatigue | 2
  Myalgia | 1
  Heat intolerance | 1
  Urethral pain | 6
  Chemical cystitis | 4
  Hematuria | 3
  Bladder spasm | 2
  Weak urinary stream | 1
  Vaginitis | 1
  Nausea | 2
  Constipation | 1
  Swelling | 4
  Pruritis | 3
  Rash | 2
  Bruising | 1
  Flushing | 1
  Dizziness | 2
  Confusion | 1
  Anxiety | 1
  Extrapyramidal symptoms | 1
  Urinary Tract Infection | 2
  Hypertension | 3

ADVERSE EVENTS:
Arm/Group | Mitomycin C With Hyperthermia
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mitomycin C With Hyperthermia (N=15)
Abdominal / pelvic discomfort (Gastrointestinal disorders) | 6 (11) — Complaint of discomfort during or post hyperthermia treatment
Bladder spasms (Renal and urinary disorders) | 2 (4)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 3 (4)
Dizziness (Nervous system disorders) | 2 (3)
Edema - localized (Blood and lymphatic system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Heat intolerance (General disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hypertension (Cardiac disorders) | 3 (7)
Induration (Skin and subcutaneous tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Urethral pain (Renal and urinary disorders) | 5 (8)
Urinary Tract Infection - suspected (Renal and urinary disorders) | 3 (3)
Vaginitis (Reproductive system and breast disorders) | 1/2 (1) — Not due to infection
constipation (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No